CLINICAL TRIAL: NCT05723406
Title: The Immunomodulatory Effect of Sugammadex After Total Hip Replacement Surgery Under Neuraxial Anaesthesia: a Pilot Study
Acronym: MAGIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL82808.091.22
Record Dates: First submitted 2023-01-27; First posted 2023-02-10 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-01

CONDITIONS: Innate Inflammatory Response; Osteoarthritis, Hip
MeSH Terms: conditions — Inflammation; Osteoarthritis, Hip | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex (Experimental): Sugammadex administration at the end of surgery
  Interventions: Drug: Sugammadex 100 MG/ML [Bridion]
- Placebo (Placebo Comparator): Placebo administration at the end of surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sugammadex 100 MG/ML [Bridion] — 8 mg/ml
  Other Names: Bridion
  Arms: Sugammadex
Other: Placebo — Sodium 0.9% 5 ml
  Arms: Placebo

SUMMARY:
Monocenter randomized controlled proof of principle study to investigate the effect of sugammadex at the end of total hip replacement surgery on the postoperative innate immune function

DETAILED DESCRIPTION:
Rationale: With infections being the number one complication after surgery, more research is aimed at therapeutic strategies that positively influence the postoperative immune dysregulation. In the search for reducing surgical stress by a deep neuromuscular block (NMB), our group recently found evidence that sugammadex, used to antagonize a deep NMB, may have an immunomodulatory effect. Ex vivo analysis showed that sugammadex counteracted the immunosuppressive effect of rocuronium, but even in absence of rocuronium it had a positive effect on cytokine production capacity.

Therefore, we now propose a clinical pilot study in patients planned for total hip surgery under neuraxial anaesthesia to further investigate whether sugammadex has beneficial immunomodulatory effects.

Primary objective: To investigate the effect of sugammadex on the postoperative innate immune function.

Study design: A blinded, randomized controlled pilot study

Study population: 20 adults scheduled for primary hip replacement surgery under neuraxial anaesthesia.

Intervention: Patients will be randomized between a group receiving sugammadex at the end of surgery and a group receiving placebo.

Primary endpoint: Postoperative innate immune function as reflected by ex vivo mononuclear cell cytokine production capacity upon whole blood lipopolysaccharide (LPS) stimulation.

Secondary endpoint: Postoperative innate immune function as reflected by DAMP release and circulating inflammatory cytokines, Quality of Recovery score (QoR-40) postoperative day 1, postoperative pain and analgesia consumption, 30-day postoperative (infectious) complications

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Scheduled for total hip replacement surgery under neuraxial anesthesia
* Scheduled for primary hip replacement surgery
* Informed consent obtained

Exclusion Criteria:

* Insufficient control of the Dutch language to read the patient information and to fill out the questionnaires
* Mentally incapacitated patients
* Known or suspected hypersensitivity to sugammadex
* Deficiency of vitamin K dependent clotting factors or coagulopathy
* Severe renal disease (creatinine clearance <30 ml/min), including patients on dialysis)
* Severe liver disease (Child-Pugh Classification C)
* Women who are or may be pregnant or currently breastfeeding
* Women of childbearing potential who don't use adequate method of contraception
* Severe vertebral column disorder
* Chronic use of psychotropic drugs
* Known hypertrophic obstructive cardiomyopathy, severe aortic valve stenosis or severe mitral valve stenosis
* Chronic use of NSAID's, steroids or immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Postoperative innate immune function | Postoperative day 1
  Ex vivo cytokine production capacity (TNF-α, IL-6, IL-10, IL-1β) of mononuclear cells upon whole blood Lipopolysaccharide(LPS) stimulation

SECONDARY OUTCOMES:
Postoperative innate immune function | 2 timepoints: At the start of surgery (±30 minutes after administration neuraxial anesthesia) and at the end of surgery (15 minutes after administration intervention/placebo medication)
  Ex vivo cytokine production capacity (TNF-α, IL-6, IL-10, IL-1β) of mononuclear cells upon whole blood Lipopolysaccharide(LPS) stimulation
Postoperative innate immune function | 3 timepoints: Postoperative day 1, at the start of surgery (±30 minutes after administration neuraxial anesthesia) and at the end of surgery (±15 minutes after administration intervention/placebo medication)
  Circulating inflammatory cytokines (TNF-α, IL-6, IL-10)
Postoperative innate immune function | 3 timepoints: Postoperative day 1, at the start of surgery (±30 minutes after administration neuraxial anesthesia), and at the end of surgery (±15 minutes after administration intervention/placebo medication)
  Danger associated molecular pattern (DAMP) release (Heat shock protein 70 (HSP 70), High mobility group box 1 (HMGB1))
Pain and total analgesia consumption | During hospital admission up to 3 days postoperative
  Pain scores by numeric rating scale (NRS 0-10)
Quality of Recovery | Postoperative day 1
  Quality of Recovery 40 (QoR-40) validated questionnaire score. 40 points (minimum: extremely poor quality of recovery) to 200 points (maximum: excellent quality of recovery)
Postoperative complications | Postoperative day 30
  postoperative complications scored by Clavien-Dindo classification; grade 0 (no deviation from ideal) grade 5 (death of patient)
Postoperative infectious complications | Postoperative day 30
  Postoperative infectious complications scored the definitions of the StEP-COMPAC group initiative

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
All data will be analyzed for publication. After that it belongs to Radboud umc where other researchers of Radboud umc may or may not include this database to their study. But there will be no active sharing

REFERENCES:
- [Derived] Bijkerk V, Jacobs LMC, Visser J, van Helden EV, Keijzer C, Helder LS, Albers KI, Warle MC. The immunomodulatory effect of sugammadex in vitro and after total hip arthroplasty : A randomised controlled pilot and retrospective cohort study. Eur J Anaesthesiol. 2025 Aug 1;42(8):676-686. doi: 10.1097/EJA.0000000000002132. Epub 2025 Feb 14. PMID 39957489
- [Derived] Jacobs LMC, Bijkerk V, van Eijk LT, Joosten LAB, Keijzer C, Visser J, Warle MC. The effect of general versus spinal anesthesia on perioperative innate immune function in patients undergoing total hip arthroplasty. BMC Anesthesiol. 2025 Jan 7;25(1):10. doi: 10.1186/s12871-024-02883-1. PMID 39773137